CLINICAL TRIAL: NCT06584773
Title: Efficacy and Impact on CMV Infection of a Quadruple Immunosuppressor Regimen With mTOR Inhibitors in Sensitized Kidney Transplant Patients
Brief Title: Efficacy of a Quadruple Immunosuppressor Regimen With mTOR Inhibitors in Sensitized Kidney Transplant Patients
Acronym: QIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Carlucci G Ventura (Unknown); Daniel R Salomon (Unknown); Fabiana Agena (Unknown); Flavio J de Paula (Unknown); Francine B Lemos (Unknown); Gislene Bezerra (Unknown); Helcio Rodrigues (Unknown); Maria da Luz Fernandes (Unknown); Nelson Zocoler Galante (Unknown); Noemia B de Lima (Unknown); Paschoalina Romano (Unknown); Patricia S Souza (Unknown); Vivian Onuchic (Unknown); Elias David Neto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE40606115.6.000.0068
Record Dates: First submitted 2024-09-02; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: kidney transplantation, sensitized, immunosuppression
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard maintenance immunosuppression (Active Comparator): tacrolimus, mycophenolate and prednisone
  Interventions: Drug: standard maintenance immunosuppression
- fourth maintenance immunosuppressive (Experimental): everolimus, tacrolimus, mycophenolate and prednisone
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — mTORi added as the fourth maintenance immunosuppressive drug in recipients
  Arms: fourth maintenance immunosuppressive
Drug: standard maintenance immunosuppression — standard maintenance immunosuppression: tacrolimus, mycophenolate, prednisone
  Arms: standard maintenance immunosuppression

SUMMARY:
In this study, sensitized renal transplant recipients, who present an increased risk of acute rejection, will be evaluated for the benefit of quadruple immunosuppression, adding sirolimus to the traditional scheme with tacrolimus, mycophenolate, and prednisone.

ELIGIBILITY:
Inclusion Criteria:

* Sensitezed renal transplant recipients with reactivity panel of antibodies (PRA) greater than 30% who agree and sign the consent form.

Exclusion Criteria:

* Obese patients (body mass index above 35 m2);
* History of GESF or membranoproliferative glomerulonephritis (MPGN) as primary cause of renal failure;
* Proteinuria (protein/creatinine ratio) greater than 0.5 mg/dL at the time of initiation of Sirolimus;
* Triglyceride levels greater than 300 mg/dl at enrollment;
* Active infection by hepatitis B virus, hepatitis C virus or HIV;
* CMV nonreactive IgG sorology at the time of transplantation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-08 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of acute rejection and/or positive viremia for CMV | From enrollment to the end of treatment at 52 weeks
  First occurrence of acute rejection and/or positive viremia for CMV, triggering early treatment within the first year after transplantation in sensitized patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Transplantation Service, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided